CLINICAL TRIAL: NCT04990973
Title: Influence of Diet on Sleep and Cardiovascular Risk
Brief Title: Evaluation of Diet and Sleep in Vascular Health: A Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot study; collection of information completed
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marie-Pierre St-Onge, Associate Professor of Nutritional Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AAAT7042; R35HL155670 (NIH)
Record Dates: First submitted 2021-07-26; First posted 2021-08-05 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Sleep
Keywords: Mediterranean diet; cardiovascular health
MeSH Terms: interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Statistician and research technicians involved in data and sample analyses will be blind to intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet and then AAD (Experimental): Healthy participants that are randomized to the MedDiet followed by a 4-week washout and a crossover to the AAD.
  Interventions: Behavioral: Average American Diet (AAD); Behavioral: Mediterranean Diet
- Average American Diet (AAD) and then Mediterranean Diet (Experimental): Healthy participants that are randomized to AAD followed by a 4-week washout and a crossover to the Mediterranean Diet.
  Interventions: Behavioral: Average American Diet (AAD); Behavioral: Mediterranean Diet

INTERVENTIONS:
Behavioral: Average American Diet (AAD) — Participants will follow specified diet requirements.
  Macronutrient targets for the AAD will be approximately 35-37% of energy from fat (13.5% from saturated fat), 15% from protein, and 48-50% from carbohydrates (10 g fiber/d for an average 2000 kcal/d diet).
Behavioral: Mediterranean Diet — Participants will follow specified diet requirements.
  Macronutrient targets for the Mediterranean diet will be approximately 40% of energy from fat (8.5% from saturated fat), 20% of energy from protein, and 40% from carbohydrates (40 g fiber/d for an average 2000 kcal/d diet).

SUMMARY:
The goal of this study is to test the impact of diet on sleep and cardiovascular disease risk factors.

DETAILED DESCRIPTION:
Poor sleep quality is highly prevalent in adults in the U.S. and worldwide. Recent work suggests that dietary intakes may influence sleep. This mechanistic study will test whether consuming a healthy, Mediterranean diet will improve sleep quality in U.S. adults with poor sleep and lead to better cardiovascular disease risk profile. Given the relationship between sleep and cardiovascular health, improving sleep quality through dietary measures could contribute to improving health in adults.

ELIGIBILITY:
Inclusion Criteria:

* Sleep >6 hours/night
* Sleep complaints

Exclusion Criteria:

* Smoking
* Allergies to foods
* Inability to comply with study procedures
* Gastrointestinal disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre St-Onge, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be shared upon request and review by investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon publication of main study outcomes.
Access Criteria: Determined upon request.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 individuals signed a consent form prior to screening assessments. Of those, 4 participants passed the eligibility criteria and were randomized to a study condition and participated in the study activities.
Groups:
- Mediterranean Diet, Then Average American Diet: Healthy participants that are randomized to the MedDiet followed by a 4-week washout and a crossover to the AAD.
  Average American Diet (AAD): Participants will follow specified diet requirements.
  Macronutrient targets for the AAD will be approximately 35-37% of energy from fat (13.5% from saturated fat), 15% from protein, and 48-50% from carbohydrates (10 g fiber/d for an average 2000 kcal/d diet).
  Mediterranean Diet: Participants will follow specified diet requirements. Macronutrient targets for the Mediterranean diet will be approximately 40% of energy from fat (8.5% from saturated fat), 20% of energy from protein, and 40% from carbohydrates (40 g fiber/d for an average 2000 kcal/d diet).
- Average American Diet, Then Mediterranean Diet: Healthy participants that are randomized to AAD followed by a 4-week washout and a crossover to the Mediterranean Diet.
  Average American Diet (AAD): Participants will follow specified diet requirements.
  Macronutrient targets for the AAD will be approximately 35-37% of energy from fat (13.5% from saturated fat), 15% from protein, and 48-50% from carbohydrates (10 g fiber/d for an average 2000 kcal/d diet).
  Mediterranean Diet: Participants will follow specified diet requirements. Macronutrient targets for the Mediterranean diet will be approximately 40% of energy from fat (8.5% from saturated fat), 20% of energy from protein, and 40% from carbohydrates (40 g fiber/d for an average 2000 kcal/d diet).
Period: First Intervention (4 Weeks)
Arm/Group | Mediterranean Diet, Then Average American Diet | Average American Diet, Then Mediterranean Diet
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Mediterranean Diet, Then Average American Diet | Average American Diet, Then Mediterranean Diet
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Mediterranean Diet, Then Average American Diet | Average American Diet, Then Mediterranean Diet
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only collected from participants who completed the study.
Groups:
- Mediterranean Diet and Then AAD: Healthy participants that are randomized to the MedDiet followed by a 4-week washout and a crossover to the AAD.
  Average American Diet (AAD): Participants will follow specified diet requirements.
  Macronutrient targets for the AAD will be approximately 35-37% of energy from fat (13.5% from saturated fat), 15% from protein, and 48-50% from carbohydrates (10 g fiber/d for an average 2000 kcal/d diet).
  Mediterranean Diet: Participants will follow specified diet requirements.
  Macronutrient targets for the Mediterranean diet will be approximately 40% of energy from fat (8.5% from saturated fat), 20% of energy from protein, and 40% from carbohydrates (40 g fiber/d for an average 2000 kcal/d diet).
- Average American Diet (AAD) and Then Mediterranean Diet: Healthy participants that are randomized to AAD followed by a 4-week washout and a crossover to the Mediterranean Diet.
  Average American Diet (AAD): Participants will follow specified diet requirements.
  Macronutrient targets for the AAD will be approximately 35-37% of energy from fat (13.5% from saturated fat), 15% from protein, and 48-50% from carbohydrates (10 g fiber/d for an average 2000 kcal/d diet).
  Mediterranean Diet: Participants will follow specified diet requirements.
  Macronutrient targets for the Mediterranean diet will be approximately 40% of energy from fat (8.5% from saturated fat), 20% of energy from protein, and 40% from carbohydrates (40 g fiber/d for an average 2000 kcal/d diet).
- Total: Total of all reporting groups
Arm/Group | Mediterranean Diet and Then AAD | Average American Diet (AAD) and Then Mediterranean Diet | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (5.7) | 34.8 (5.7) | 34.8 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 2 | 2
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4
PSQI [Mean (Standard Deviation); unit: units on a scale] | 3.5 (0.7) | 5 (1.4) | 4.3 (1.3)
Sleep Fragmentation Index [Mean (Standard Deviation); unit: percent] — Sleep Fragmentation is an index of restlessness during the sleep period expressed as a percentage (0 to 100%). The higher the index, the more sleep is disrupted. Two weeks prior to randomization, participants will wear an actigraph monitor and keep a sleep diary to verify sleep duration and quality.
  percent | 29.9 (8.9) | 15.9 (5.5) | 22.9 (10.1)
Sleep duration [Mean (Standard Deviation); unit: minutes per night] — Sleep duration reported as average amount of sleep (in minutes) per night. Two weeks prior to randomization, participants will wear an actigraph monitor and keep a sleep diary to verify sleep duration and quality.
  minutes per night | 386.6 (17.0) | 402.4 (26.2) | 394.5 (20.2)

OUTCOME MEASURES:

1. Primary Outcome: Score on the Pittsburgh Sleep Quality Index (PSQI)
Description: The 19 questions which compose this survey assess sleep quality, latency, duration, habitual sleep efficiency, sleep disturbances, medication use and daytime dysfunction. Scores range 0 (minimum) to 21 (maximum) with >5 indicating poor sleep quality so a lower score is a better outcome.
Time Frame: 4 weeks
Population: 1 participant in the Mediterranean Diet condition did not complete the questionnaire.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mediterranean Diet Condition: Mediterranean Diet: Participants will follow specified diet requirements.
  Macronutrient targets for the Mediterranean diet will be approximately 40% of energy from fat (8.5% from saturated fat), 20% of energy from protein, and 40% from carbohydrates (40 g fiber/d for an average 2000 kcal/d diet).
- Average American Diet (AAD) Condition: Average American Diet (AAD): Participants will follow specified diet requirements.
  Macronutrient targets for the AAD will be approximately 35-37% of energy from fat (13.5% from saturated fat), 15% from protein, and 48-50% from carbohydrates (10 g fiber/d for an average 2000 kcal/d diet).
Arm/Group | Mediterranean Diet Condition | Average American Diet (AAD) Condition
Number analyzed (Participants) | 3 | 4
units on a scale | 0.3 (1.5) | -0.5 (2.1)

2. Primary Outcome: Sleep Fragmentation Index
Description: Sleep Fragmentation is an index of restlessness during the sleep period expressed as a percentage (0 to 100%). The higher the index, the more sleep is disrupted.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Mediterranean Diet: Macronutrient targets for the Mediterranean diet will be approximately 40% of energy from fat (8.5% from saturated fat), 20% of energy from protein, and 40% from carbohydrates (40 g fiber/d for an average 2000 kcal/d diet).
- Average American Diet (AAD): Macronutrient targets for the AAD will be approximately 35-37% of energy from fat (13.5% from saturated fat), 15% from protein, and 48-50% from carbohydrates (10 g fiber/d for an average 2000 kcal/d diet).
Arm/Group | Mediterranean Diet | Average American Diet (AAD)
Number analyzed (Participants) | 4 | 4
percent | 11.0 (2.8) | 15.8 (8.4)

3. Primary Outcome: Average Sleep Duration Per Night
Description: Sleep duration will be actigraphy-derived.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: minutes per night
Arm/Group | Mediterranean Diet | Average American Diet (AAD)
Number analyzed (Participants) | 4 | 4
minutes per night | 403.7 (52.0) | 424.0 (51.3)

4. Secondary Outcome: Change in Urinary 6-sulfatoxymelatonin Level
Description: Urinary 6-sulfatoxymelatonin will be measured by competitive ELISA and urine creatinine by clinical chemistry analyzer.
Time Frame: Change from baseline to 4 weeks
Population: Due to study termination, data was not collected and therefore not analyzed.
Arm/Group | Mediterranean Diet | Average American Diet (AAD)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Tryptophan
Description: Tryptophan metabolism
Time Frame: Change from baseline to 4 weeks
Population: Due to study termination, data was not collected and therefore not analyzed.
Arm/Group | Mediterranean Diet | Average American Diet (AAD)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Kynurenine
Description: Tryptophan metabolism
Time Frame: Change from baseline to 4 weeks
Population: Due to study termination, data was not collected and therefore not analyzed.
Arm/Group | Mediterranean Diet | Average American Diet (AAD)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Serotonin
Description: Neurotransmitter
Time Frame: Change from baseline to 4 weeks
Population: Due to study termination, data was not collected and therefore not analyzed.
Arm/Group | Mediterranean Diet | Average American Diet (AAD)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study intervention timeframe (approximately 12 weeks)
Groups:
- Mediterranean Diet: Healthy participants that are randomized to the MedDiet followed by a 4-week washout and a crossover to the AAD.
  Average American Diet (AAD): Participants will follow specified diet requirements.
  Macronutrient targets for the AAD will be approximately 35-37% of energy from fat (13.5% from saturated fat), 15% from protein, and 48-50% from carbohydrates (10 g fiber/d for an average 2000 kcal/d diet).
  Mediterranean Diet: Participants will follow specified diet requirements.
  Macronutrient targets for the Mediterranean diet will be approximately 40% of energy from fat (8.5% from saturated fat), 20% of energy from protein, and 40% from carbohydrates (40 g fiber/d for an average 2000 kcal/d diet).
- Average American Diet (AAD): Healthy participants that are randomized to AAD followed by a 4-week washout and a crossover to the Mediterranean Diet.
  Average American Diet (AAD): Participants will follow specified diet requirements.
  Macronutrient targets for the AAD will be approximately 35-37% of energy from fat (13.5% from saturated fat), 15% from protein, and 48-50% from carbohydrates (10 g fiber/d for an average 2000 kcal/d diet).
  Mediterranean Diet: Participants will follow specified diet requirements.
  Macronutrient targets for the Mediterranean diet will be approximately 40% of energy from fat (8.5% from saturated fat), 20% of energy from protein, and 40% from carbohydrates (40 g fiber/d for an average 2000 kcal/d diet).
Arm/Group | Mediterranean Diet | Average American Diet (AAD)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT04990973/Prot_SAP_000.pdf